CLINICAL TRIAL: NCT03600519
Title: Retinal Imaging Using NOTAL-OCT V2.5
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: BNZ-0060-18
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: AMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMD Patients: OCT scan
  Interventions: Device: NOTAL OCT V2.5

INTERVENTIONS:
Device: NOTAL OCT V2.5 — AMD Patients
  Other Names: OCT scan

SUMMARY:
Primary objectives:

To compare between retinal measurements, done by the NOTAL-OCT V2.5 device and a commercial OCT.

Secondary objectives:

1. To evaluate the level of agreement between the NOTAL-OCT V2.5 and a commercial OCT in the presence of fluid as identified in the OCT images, in the central 10 degrees of the macula.
2. To evaluate the repeatability of the NOTAL-OCT V2.5

DETAILED DESCRIPTION:
Study population:

1. AMD population - intermediate and advanced AMD (with active and nonactive CNV)
2. DR population. Patient with and without DME

ELIGIBILITY:
1. Inclusion Criteria:

   a- Ability and agreement to give informed consent (IC) b -Diagnosis of AMD or DR in SE by OCT c- Ability to undergo OCT scans d- VA of 20/400 (6/120) or better in SE
2. Exclusion Criteria:

   1. AMD and DR in the same SE
   2. Evidence of macular disease other than AMD or DME in SE
   3. Patient with dilated eye(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MAD patients
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-07-22 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The level of agreement between NOTAL-OCT V2.5 and commercial OCT in detecting fluid | less than an hour
  measurements of retinal thickness.

CONTACTS AND LOCATIONS:
Locations (1):
- Bnei Zion, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided